CLINICAL TRIAL: NCT02086539
Title: A Randomized Controlled Trial of Outreach Approaches to Increase Enrollment in the Habit Formation for Adherence to Statin Use and LDL Reduction Study
Brief Title: Comparison of Outreach Approaches to Increase Enrollment in a Healthy Cholesterol Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Rutgers University (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 816003; 5R01AG043844-02 (NIH)
Record Dates: First submitted 2014-03-11; First posted 2014-03-13 (Estimated); Last update posted 2017-06-27 (Actual); Status verified 2017-06

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Normal Letter (No Intervention): This arm will receive the recruitment letter in a business sized envelope. The letter states the participant will receive a $25 check upon enrollment into the study.
- Large Envelope (Experimental): This arm will receive the recruitment letter in an 8.5 x 11 inch envelope. The letter states the participant will receive a $25 check upon enrollment into the study.
  Interventions: Other: Large Envelope
- Priority Mail (Experimental): Group 3 will receive a recruitment letter shipped via USPS priority mail. The letter states the participant will receive a $25 check upon enrollment into the study.
  Interventions: Other: Priority Mail
- Amazon (Experimental): This arm will receive a recruitment letter with the image of an Amazon gift card and told they will receive the $25 gift card if they enroll in the study.
  Interventions: Other: Amazon

INTERVENTIONS:
Other: Large Envelope
  Arms: Large Envelope
Other: Priority Mail
  Arms: Priority Mail
Other: Amazon
  Arms: Amazon

SUMMARY:
This study aims to determine the effectiveness of 4 different recruitment techniques for enrollment into a cholesterol study. 2,000 people that meet initial eligibility criteria for the study will be randomized into one of 4 groups and will all receive the same recruitment letter inviting them to participate in the study by enrolling on an online platform. Group 1 will receive the recruitment letter in a normal sized envelope, Group 2 will receive the recruitment letter in an 8.5 x 11 inch envelope, Group 3 will receive a recruitment letter shipped via USPS priority mail and a Group 4 will receive a recruitment letter with the image of an Amazon gift card and told they will receive a $25 gift card if they enroll in the study. All other groups are told that they will receive a $25 check upon enrollment in the study.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes and or history of CVD
* LDL > or = 130 mg/dl - measured during screening
* A prescription filled for statin medication within the last 12 months
* Medication Possession Ratio (MPR) <80%
* CVS Caremark Beneficiary

Exclusion Criteria:

* Less than 18 years old
* Contraindication to further statin use or have suffered side effects from statins, such as myopathy
* Will not or cannot give consent
* History of active or progressive liver disease or abnormal liver function tests on baseline screening
* Currently participating in another clinical trial with related aims
* Co-morbidities likely to lead to death within a short-period

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-04; Primary Completion 2016-07-23 (Actual); Study Completion 2016-07-23 (Actual)

PRIMARY OUTCOMES:
Enrollment into the Habit Formation study | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Kevin G Volpp, MD, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States